CLINICAL TRIAL: NCT00315471
Title: VCRC Longitudinal Protocol for Takayasu's Arteritis
Brief Title: Determining Disease Activity Biomarkers in Individuals With Takayasu's Arteritis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Principal Investigator, Peter Merkel, Professor, University of Pennsylvania
Other Study IDs: VCRC5503; U54AR057319 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Takayasu's Arteritis
Keywords: Vasculitis
MeSH Terms: conditions — Takayasu Arteritis; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum and plasma), urine, and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Takayasu's arteritis is a rare disorder that causes swelling and damage to the large arteries in the body, such as the aorta. In order to ensure proper treatment, measuring disease activity is critical. The purpose of this study is to establish new biological markers (biomarkers) to assess the severity of disease in people with Takayasu's arteritis.

DETAILED DESCRIPTION:
Takayasu's arteritis is a chronic inflammatory condition that affects the aorta, the largest blood vessel in the body, and its branches. Inflammation causes segments of the vessels to become narrowed, blocked, or even stretched, possibly resulting in aneurysms. The disease is very rare but most commonly occurs in young Asian women. Symptoms may include arm pain with use, decreased or absent pulses, lightheadedness or dizziness, headaches, and visual disturbances. Many individuals with Takayasu' arteritis, however, have no apparent symptoms despite disease activity. Additionally, current tests used to measure vessel inflammation are considered unreliable and inconsistent. It is therefore very difficult to determine the extent of disease activity in a person with Takayasu's arteritis. This study will use novel scientific methods to establish new biomarkers that can be used to monitor disease activity in individuals with Takayasu's arteritis. These biomarkers may be used to help direct clinical care and assist in future drug development.

Study visits will occur monthly for the first year, then every 3 months thereafter for the remainder of the study. Blood and urine collection will occur at every visit. A physical examination, disease assessment, and review of medications will occur every 3 months; participants may also be asked to complete various questionnaires. Diagnostic testing, which may include chest radiograph, echocardiogram, magnetic resonance imaging, or angiography, will occur every 6 months. Tobacco, alcohol, and drug use will be assessed on a yearly basis. Participants may have additional study visits if a disease flare or disease-related complications occur during the study.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of arteriogram abnormalities compatible with Takayasu's arteritis (includes conventional dye angiography, magnetic resonance angiography, or computed tomography angiography)
* Evidence of one of the following criteria:

  1. Age at disease onset of 50 years or younger
  2. Claudication of the arms or legs
  3. Decreased brachial artery pulse (one or both arteries)
  4. Blood pressure difference between the arms of at least 10 mm Hg
  5. Bruit over the subclavian arteries or aorta
* Parental consent for children under the age of 18

Exclusion Criteria:

* Arteriographic lesions that could be entirely due to atherosclerosis
* Fibromuscular dysplasia
* Cogan's syndrome
* Behcet's disease
* Sarcoidosis
* Kawasaki disease
* Giant cell arteritis (large vessel vasculitis and at least 50 years old)
* Syphilis or other infectious forms of large vessel vasculitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Takayasu's arteritis. Enrollment will be sequential and participants will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Discover biomarkers in Takayasu's arteritis capable of measuring disease activity and response to treatment. | Study completion

SECONDARY OUTCOMES:
Measure the predictive value of biomarkers for clinical outcome in Takayasu's arteritis. | Study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Merkel, MD, MPH, Study Director — Vasculitis Clinical Research Consortium (VCRC)
Locations (9):
- United States (7):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sueyoshi E, Sakamoto I, Ogawa Y, Uetani M. Diagnosis of perfusion abnormality of the pulmonary artery in Takayasu's arteritis using contrast-enhanced MR perfusion imaging. Eur Radiol. 2006 Jul;16(7):1551-6. doi: 10.1007/s00330-005-0095-z. Epub 2006 Jan 14. PMID 16416104
- [Background] Ng WF, Fantin F, Ng C, Dockery F, Schiff R, Davies KA, Rajkumar C, Mason JC. Takayasu's arteritis: a cause of prolonged arterial stiffness. Rheumatology (Oxford). 2006 Jun;45(6):741-5. doi: 10.1093/rheumatology/kei274. Epub 2006 Jan 10. PMID 16403827
- [Background] Park MC, Lee SW, Park YB, Lee SK. Serum cytokine profiles and their correlations with disease activity in Takayasu's arteritis. Rheumatology (Oxford). 2006 May;45(5):545-8. doi: 10.1093/rheumatology/kei266. Epub 2005 Dec 13. PMID 16352633
- [Background] Tripathy NK, Gupta PC, Nityanand S. High TNF-alpha and low IL-2 producing T cells characterize active disease in Takayasu's arteritis. Clin Immunol. 2006 Feb-Mar;118(2-3):154-8. doi: 10.1016/j.clim.2005.09.010. Epub 2005 Dec 7. PMID 16337833
- [Background] Park MC, Lee SW, Park YB, Chung NS, Lee SK. Clinical characteristics and outcomes of Takayasu's arteritis: analysis of 108 patients using standardized criteria for diagnosis, activity assessment, and angiographic classification. Scand J Rheumatol. 2005 Jul-Aug;34(4):284-92. doi: 10.1080/03009740510026526. PMID 16195161
- See also: Vasculitis Clinical Research Consortium — http://rarediseasesnetwork.org/cms/vcrc
- See also: Rare Diseases Clinical Research Network — http://rarediseasesnetwork.org